CLINICAL TRIAL: NCT05506553
Title: A Randomised, Controlled Study to Compare Visual Performance Following Bilateral, Micro-monovision Insertion of Two Toric, Aspheric, Hydrophobic Acrylic Intraocular Lenses: The TECNIS Eyhance Toric II IOL and the Alcon Acrysof IQ Toric IOL
Brief Title: Comparison of Aspheric Toric Intraocular Lenses for Micro-monovision
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: City, University of London (Other); King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 311123
Record Dates: First submitted 2022-07-14; First posted 2022-08-18 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-07

CONDITIONS: Cataract; Presbyopia; Astigmatism
Keywords: Cataract; Presbyopia; Astigmatism
MeSH Terms: conditions — Cataract; Presbyopia; Astigmatism | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Randomised Control Trial
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Control arm (Active Comparator): Bilateral insertion of Alcon IQ Toric IOL in micro-monovision
  Interventions: Device: Control Arm - Alcon IQ Toric Intraocular lens
- Intervention arm (Experimental): Bilateral insertion of Eyhance Toric II IOL
  Interventions: Device: Intervention arm - Eyhance Toric II Intraocular Lens

INTERVENTIONS:
Device: Intervention arm - Eyhance Toric II Intraocular Lens — Bilateral cataract extraction and insertion of Eyhance Toric II Intraocular Lens
  Arms: Intervention arm
Device: Control Arm - Alcon IQ Toric Intraocular lens — Bilateral cataract extraction and insertion of Alcon IQ Toric Intraocular Lens
  Other Names: Control Group
  Arms: Control arm

SUMMARY:
In an aging population, cataract and presbyopia become increasingly common. A cataract is the opacification of the natural crystalline lens inside a person's eye, causing reduction of vision. Presbyopia is an age related condition resulting in loss of reading/near vision which results in requiring reading glasses.

Astigmatism is a common condition characterized by an abnormal cornea (the clear tissue at the front of the eye) which results in blurred distance and near vision, again requiring glasses.

Cataract surgery is the most common elective surgery worldwide for patients over 65. It is composed of removal the cataract and insertion of a new intraocular lens (IOL). Currently only monofocal IOLs are available on the National Health Service (United Kingdom) - meaning they give good distance or near vision. The majority of patients opt for good distance vision with glasses to read.

The investigators are trialling insertion of a new Extended Depth of Focus (enhanced aspheric) Toric IOL (EDoF Toric IOL), which treats all 3 conditions - cataract, presbyopia and astigmatism. All patients attending St Thomas' hospital for treatment of cataracts, who have presbyopia and astigmatism will be considered for invitation to the study.

Patients who participate in the study will be randomly selected to receive either the new IOL - the TECNIS Eyhance Toric II IOL, or a well-established IOL the Alcon Acrysof IQ Toric IOL during cataract surgery. Insertion of the Alcon Acrysof IQ Toric IOL is known to treat cataract and astigmatism but not presbyopia.

Patients will be assessed and have their surgery performed at St Thomas' Hospital London. They will have 7 appointments over 12 months, plus surgery. The investigators hope to demonstrate better distance, intermediate and near vision and increased spectacle independence in the TECNIS Eyhance Toric II IOL group.

EDoF Toric IOLs have the potential to transform cataract surgery outcomes for patients in the NHS.

DETAILED DESCRIPTION:
Cataract is a condition caused by progressive clouding of the natural crystalline lens inside the eye. This leads to impairment of visual performance. This condition represents a huge disease burden and is a leading cause of reversible blindness worldwide. In the UK and the developed world, the incidence of cataract induced blindness continues to increase, secondary to an aging population and increasingly common risk factors such as diabetes. In 1950, Harold Ridley inserted an intraocular lens following cataract extraction at St Thomas' Hospital. This was the first recorded surgery of its kind, and heralded the development of modern cataract surgery, which is comprised of extraction of a cataract by phacoemulsification (ultrasonic micro-fragmentation) followed by insertion of a foldable intraocular lens. Cataract surgery (CS) is the most common elective surgical procedure in the developed world, and the most common in the EU, with 4 million procedures performed in 2016. CS continues to evolve, as do intraocular lenses (IOLs).

Currently, only mono-focal (one point of focus) IOLs are available during cataract surgery in the NHS. These are designed to give excellent vision for one fixed point of focus (either distance, intermediate or near vision), with most patients opting for good distance vision, and requiring glasses for intermediate vision or near vision. Accordingly, these lenses do not treat presbyopia, the loss of the ability focus on near objects, that most people develop in their 50's. In addition, the standard monofocal lens does not treat astigmatism, a common condition characterized by a non-spherically shaped cornea (the clear tissue at the front of the eye) which results in blurred unaided distance and near vision and the need for both reading and distance glasses following surgery.

In this trial patients will be randomly assigned to receive two TECNIS Eyhance Toric lenses or two Alcon Acrysof IQ Toric II lenses (one for each eye). Prior to surgery the 'power' of each patients intraocular lens is chosen. This is similar to choosing the power of lenses in spectacles at an opticians. By choosing the power of one eye to be targeted for distance and the other offset for a small myopic (short-sighted) correction to allow unaided intermediate (computer) and some unaided near vision, the investigators can then investigate the efficacy of these lenses not only to improve vision after cataract surgery but also their ability to treat astigmatism and reduce the dependence on spectacles following NHS CS. As such the investigators hope to offer cost benefits to NHS patients as well as quality of life improvements. In addition to efficacy, quality of life and cost benefits to patients, the investigators will also explore patient acceptability of such "premium" IOLs and look at models to investigate their affordability with the NHS setting.

This study is a clinical trial, designed to compare visual outcomes after cataract surgery with two different intraocular lenses. As previously described, modern day cataract surgery is composed of two main components: removal of the cataract, and insertion of an intraocular lens (IOL). The role of the intraocular lens is to replace the focusing power of the natural crystalline lens inside the eye. It is this lens that becomes a cataract. Removing a cataract alone helps light enter the eye, but does not focus it well. Prior to the invention of intraocular lenses, patients required extremely thick and strong glasses for both distance vision.

Currently only monofocal intraocular lenses are available on the NHS. Different strengths of lens can be chosen to give the patient good distance, intermediate or near vision. That means the ability to focus on objects in the distance, middle distance or near. Most patients opt for good distance vision, enabling them to mobilise easily, watch TV and drive, and require glasses for reading.

As described above, most patients over the age of 50, have some element of presbyopia, which is the inability to focus on near objects, resulting in the need for reading glasses. Inserting extended depth of focus (EDoF IOLs) intraocular lenses during cataract surgery, can help improve their reading vision without reading glasses.

Astigmatism is an abnormality of the cornea, which requires special distance and reading glasses to give clear distance and near vision. Toric IOLs correct astigmatism and reduce or prevent the need for astigmatism correcting glasses after surgery.

The TECNIS Eyhance Toric II IOL is a new IOL which corrects astigmatism and has an enhanced depth of focus through its novel 'enhanced aspheric' design. This will help treat presbyopia. The Alcon Acrysof IQ Toric IOL is an established Toric IOL corrects astigmatism alone.

This trial will investigate the effect of a new Extended depth of focus (enhanced aspheric) toric lens on vision and compare it to a commonly used Toric IOL. The investigators will recruit patients who have bilateral cataracts with astigmatism. These patients will have otherwise healthy eyes. Patients who have been referred to St Thomas' Hospital for assessment for cataracts will be considered for the trial. If they fulfil the criteria for acceptance to the trial, the consulting doctor will discuss this with the patient. If the patient expresses interest, they will be referred to the Research department. The cataract research fellow will review them and consider them for admission to the trial. This review will happen on the day of the original appointment, or the patient will be given an another appointment time and date for further assessment. If a patient would like further information about the study, but cannot speak to the Cataract Research Fellow that same day, they will be asked to fill in a Consent to Contact form, which will allow the research department to contact the patient for consideration for entry to the study.

The investigators will recruit 2 groups of patients, with 70 patients in each group. The investigators will randomly assign them to either the TECNIS Eyhance Toric II group or the Alcon Acrysof IQ Toric IOL group. All patients will cataract surgery on one eye, appointments to review their progress, and then the second cataract operation. The patients in the TECNIS Eyhance group will have TECNIS Eyhance Toric II lenses inserted into both eyes. The patients in the Alcon Acrysof IQ Toric group will have Alcon Acrysof Toric IQ lenses inserted into both eyes. Patients who fulfil the inclusion/exclusion criteria will be fully informed of the investigative nature of the study and consented. Neither the TECNIS Eyhance Toric II IOL or the Alcon Acrysof IQ Toric IOL are used in the NHS, but are used in private practice in the UK

Once patients are consented, they will have a pre-operative assessment which will include a full eye examination (including biomicroscopy and tonometry), refraction (a glasses similar to a visit to an opticians), have their vision tested at near, intermediate and distance with and without glasses. They will also have contrast sensitivity (previously described), pentacam scanning (mapping of the front of the eye) and an intraocular pressure check. The investigators will perform a biometry (measurement of the eye) to calculate the lens power required for surgery. Intraocular lenses are available in different powers, in the same way spectacle lenses are available in different powers.

Cataract surgery will be performed during National Health Service (United Kingdom) cataract lists at St Thomas' Hospital. Surgery will be performed by senior cataract surgeons, and standard protocols will be followed. Patients will be reviewed at 2 weeks, 6 weeks and 6 months after surgery.

The 2 weeks post operative review will be collect the same data as the pre-operative assessment as described above. Patients reviewed at 6 week and 6 months post operation will have all of the above, plus digital imaging (photography), stereoacuity (3d vision) and ScheimpflugTomography (3d scanning) to assess IOL tilt and decentration. The digital photography will be compared with a digital photograph taken on the day of surgery, to assess rotational lens stability. The 6 month digital image will be used to assess posterior capsular opacification and glistenings (problems with the lens or behind the lens). Anonymised digital images may be shared with Prof Chris Hull at City University to help us assess glistening of the IOLs. At pre-operative assessment and 6 week assessment a scan of the macula (macula OCT) will take place. This is a noninvasive test done in the eye department.

Participants in the study at the 6 weeks-, 6-month visits should expect to take around an extra 120 minutes in total for these extra, non-invasive tests to be performed. Patients will be asked to complete questionnaires, namely EQ-5D-3L, Catquest-9SF and Cat-PROM, before surgery- and at 6 week and 6 months post-operatively. At 6 months, the need for, type of and expenditure cost of spectacles required by patients will be recorded and compared between groups. Finally patients will be monitored for adverse events at every appointment after surgery.

Interim data will be reviewed at 20% completion of treatment and 6 month followup (following second eye surgery). The study completion date will be when Patient 140 has completed their 6 month visit (following second eye surgery) plus 14 days for data entry and database lock.

The investigators will be using a strategy called micro-monovision. Most people have a dominant eye, in the same way that they have a dominant hand. In micro-monovision the investigators choose an intraocular lens power that will give the dominant eye good distance vision (emmetropia), and a intraocular lens power that will give the non-dominant eye good intermediate distance vision. The investigators will be using this strategy in both the TECNIS Eyhance Toric II group and the Alcon IQ Toric group.

The investigators are testing the following hypotheses (theories)

1. That the TECNIS Eyhance Toric IOL, when implanted in both eyes, will give better middle distance and near vision, than the Alcon IQ Toric lens, whilst maintaining a similarly good quality of good distance vision. The investigators will also compare contrast sensitivity and stereoacuity (described previously). The investigators will also record complaints of 'flashing lights' or 'halos' in a patients vision, which can be caused by the implantation of the intraocular lens. These are considered to be a rare side effect.
2. That the TECNIS Eyhance Toric II IOL, when implanted in both eyes, will give better middle distance and near vision, than the Alcon Acrysof IQ Toric lens, resulting in improved patient satisfaction scores on the CatPROM and CatQUEST trial.
3. That the TECNIS Eyhance Toric II IOL, when implanted in both eyes, will give better middle distance and near vision, than the Alcon Acrysof IQ Toric lens, thus resulting in reduced costs for the patient, as they will not need to buy reading or intermediate vision glasses.
4. That the TECNIS Eyhance Toric II IOL, when implanted in both eyes, will give better middle distance and near vision, than the Alcon Acrysof IQ Toric lens, has similar stability, and does not rotate.

ELIGIBILITY:
Inclusion Criteria:

* Bilateral cataract requiring surgical intervention,
* age over 18 years
* able to understand informed consent and the objectives of the trial,
* not pregnant, not breast feeding
* no previous intraocular eye surgery
* good visual potential in both eyes
* corneal astigmatism of 1.5 to 6 dioptres

Exclusion Criteria:

* Any patient with other ocular condition that might reduce visual acuity and hence confound the results such as:
* visually impairing age-related macular degeneration
* Advanced glaucoma
* previous retinal vascular disorders
* previous retinal detachment or tear
* any visually impairing neuro-ophthalmological condition
* any inherited retinal disorder or pathology
* previous strabismus surgery or record of amblyopia
* previous visually impairing CVA, TIA or other vaso-occlusive disease
* already enrolled in another study or trial
* instability of keratometry or biometry measurements
* irregular astigmatism
* previous significant trauma to eye

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Change in Refractive Error from baseline to 6 weeks | 6 weeks after cataract surgery
  Optometrist assessed refractive error for Near, and distance vision
Change in Refractive Error from baseline to 6 months | 6 months after cataract surgery
  Optometrist assessed refractive error for Near, and distance vision
Change in Visual acuity from baseline to 6 weeks | 6 weeks after each cataract surgery
  Uniocular - unaided and best corrected near, intermediate and distance vision Binocular - unaided and best corrected near, intermediate and distance vision
Change in Visual acuity from baseline to 6 months | 6 months after each cataract surgery
  Uniocular - unaided and best corrected near, intermediate and distance vision Binocular - unaided and best corrected near, intermediate and distance vision
Change in Patient Satisfaction from baseline to 6 weeks | 6 weeks after each cataract surgery
  Patient satisfaction - PROM questionnaire EQ-5D-3L
Change in Patient Satisfaction from baseline to 6 weeks | 6 weeks after each cataract surgery
  Patient satisfaction - PROM questionnaire Catquest-9SF
Change in Patient Satisfaction from baseline to 6 weeks | 6 weeks after each cataract surgery
  Patient satisfaction - PROM questionnaire Cat-PROM
Change in Patient Satisfaction from baseline to 6 months | 6 months after each cataract surgery
  Patient satisfaction - PROM questionnaire EQ-5D-3L
Change in Patient Satisfaction from baseline to 6 months | 6 months after each cataract surgery
  Patient satisfaction - PROM questionnaire Catquest-9SF
Change in Patient Satisfaction from baseline to 6 months | 6 months after each cataract surgery
  Patient satisfaction - PROM questionnaire Cat-PROM
Change in rotational stability of Intraocular lens relative to its intended angle of insertion from baseline to 6 weeks | 6 weeks after each cataract surgery
  IOL rotation judged using colour photography
Change in rotational stability of Intraocular lens relative to its intended angle of insertion from baseline to 6 months | 6 months after each cataract surgery
  IOL rotation judged using colour photography
Patient related cost benefits in terms of spectacle expenditure. | 6 months after second eye cataract surgery
  Cost of spectacles purchased after cataract surgery will be compared between the two group

SECONDARY OUTCOMES:
Change in Stereoacuity at 6 weeks after second eye surgery | 6 weeks after second cataract surgery
  Randot stereoacuity test
Change in Stereoacuity at 6 months after second eye surgery | 6 months after second cataract surgery
  Randot stereoacuity test
Change in Contrast sensitivity at 6 weeks after cataract surgery | 6 weeks after each cataract surgery
  CSV-1000
Change in Contrast sensitivity at 6 months after cataract surgery | 6 months after each cataract surgery
  CSV-1000
Post-operative complications 2 weeks after surgery | 2 weeks after each cataract surgery
  Documentation of post-operative complications, including extent of Posterior Capsular Opacification and lens glistenings on digital imaging
Post-operative complications 6 weeks after surgery | 6 weeks after each cataract surgery
  Documentation of post-operative complications, including extent of Posterior Capsular Opacification and lens glistenings on digital imaging
Post-operative complications 6 months after surgery | 6 months after each cataract surgery
  Documentation of post-operative complications, including extent of Posterior Capsular Opacification and lens glistenings on digital imaging
Change in IOL decentration and tilt seen on Scheimpflug tomography (Pentacam) at 6 weeks | 6 weeks after each cataract surgery
  IOL decentration and tilt seen on Scheimpflug tomography (Pentacam)
Change in IOL decentration and tilt seen on Scheimpflug tomography (Pentacam) at 6 months | 6 months after each cataract surgery
  IOL decentration and tilt seen on Scheimpflug tomography (Pentacam)

CONTACTS AND LOCATIONS:
Overall Officials: David O'Brart, MBBS, MD, Study Director — Guy's and St Thomas' NHS Foundation Trust
Locations (1):
- St Thomas' Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No